CLINICAL TRIAL: NCT05321680
Title: Withdrawal of Antidementia Drugs in Advanced Dementia (WADAD): a Randomized Clinical Trial and Cost-utility Analysis
Brief Title: Withdrawal of Antidementia Drugs in Advanced Dementia (WADAD)
Acronym: WADAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Veronica Raquel Alheia Cabreira, Principal Investigator, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68-21
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Dementia
Keywords: antidementia drug; dementia; quality of life; cost-utility analysis
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A clinical, pragmatic, unicentric, open trial with blinded assessors. We will use a parallel randomized design (1:1) that will evaluate the effect of maintaining pharmacological treatment versus treatment withdrawal.
Who Masked: Outcomes Assessor
Masking Description: anonimized data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment withdrawal (Experimental): discontinuation of treatment (anti-cholinesterase inhibitors including donepezil, rivastigmine and galantamine; and/or memantine)
  Interventions: Other: Treatment withdrawal
- Treatment continuation (No Intervention): treatment continuation (anti-cholinesterase inhibitors including donepezil, rivastigmine and galantamine; and/or memantine)

INTERVENTIONS:
Other: Treatment withdrawal — Tapering or suspension of antidementia drugs
  Arms: Treatment withdrawal

SUMMARY:
Dementia is a chronic progressive mental disorder that adversely affects higher cortical functions, including cognition and behavior leading up to disability and dependence in daily life activities. It has become a major public health concern because of its increasing prevalence, chronicity, burden for caregivers, and the high personal and financial costs needed for care. Alzheimer disease (AD) is the most prevalent form of dementia, occurring in 5% to 7% of individuals older than 60. In Portugal, Santana et al study estimated that 160 287 people above 60 years had a diagnosis of dementia in 2013 (prevalence of 5,9%).The increasing national and international prevalence of dementia and its associated burden then imparts a high priority on delivering safe and effective treatment options.

Currently approved treatments available for the symptomatic management of mild to moderate AD include cholinesterase inhibitors (ChEIs) (donepezil, rivastigmine, and galantamine) and a N-methyl- D-aspartate receptor antagonist (memantine). These drugs are also given off-label for other types of dementia (vascular and mixed dementias), with treatment continuing through advanced disease stages. Given that ChEIs have demonstrated short-term modest stabilization on measures of cognition and global functioning in randomized controlled trials (RCTs), several practice guidelines have proposed ChEIs for the treatment of all stages of AD, with some advocating ChEI discontinuation if tolerability issues arise, or if there is no longer a noticeable clinical benefit. Further studies in this setting are important as patients with severe dementia are more functionally impaired, present with comorbid illnesses, posing a higher risk of polypharmacy. In addition, ChEIs have a potential risk of adverse events including nausea, diarrhea, insomnia, vomiting, muscle cramping, fatigue, and weight loss. Less commonly, ChEI might be associated with rhabdomyolysis, convulsions, falls, syncope, pneumonia and death. Because cognitive and behavioral impairments change during the progressive disease course, the effects of medications may be unpredictable, especially over long durations of treatment. It might be challenging to weigh minimally beneficial effects against predicted harms of continued treatment, considering both patient and caregiver-centered care goals besides less clinically relevant cognitive outcomes.

Only a small number of discontinuation RCTs were conducted to date but involved relatively few participants with heterogeneous designs, disease severities and outcomes. As so, clinicians take individualized discontinuation decisions and the only consensual domains are a lack of response and a loss of effectiveness. The present pragmatic clinical trial will compare the efficacy of maintaining pharmacological treatment versus treatment cessation on cognition, behavior, functional disability and quality of life of patients and caregivers, among patients with severe dementia due to AD, with or without small vessel subcortical vascular disease. The investigators will consider other important endpoints besides cognitive functioning including mood, apathy, energy and neuropsychiatric symptoms. Moreover, this trial will try to look for outcomes that engage patients and families in treatment decisions.

DETAILED DESCRIPTION:
Specific aim 1. Explore the effects of discontinuing ChEI and/or memantine on global impression, disease severity, function, behavior and cognitive outcomes;

Hypothesis:

1. Progression to disability (defined as a loss of 2 of 4 basic functions, or 6 of 11 instrumental functions, according to the BADLS), at 6 months, is significantly higher in patients discontinuing therapy;
2. Patients with severe dementia who discontinue ChEI and/or memantine show a significantly higher decline on ratings of cognitive function, behavior and activities of daily living over 6 months than those continuing these drugs;
3. Patients with severe dementia who discontinue ChEI and/or memantine experience increased adverse events including healthcare visits and other several medical intercurrences.

Specific aim 2. Explore the effects of discontinuation strategies in patients and caregiver's health related quality of life.

Hypothesis:

a) Patients with severe dementia and their caregivers experience lower levels of health-related quality of life after treatment discontinuation.

Specific aim 3. Cost-utility and cost-effectiveness analysis of a discontinuation strategy.

a) Treatment with antidementia drugs is the most cost-effective treatment strategy in advanced stages of dementia, delaying progression to disability and reducing formal and informal costs and healthcare utilization;

a) Treatment with antidementia drugs is the strategy associated with better quality of life and lower cost-utility ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of dementia syndrome defined by clinical criteria (Alzheimer's dementia according to NIA-AA 2011 criteria, vascular dementia or mixed dementia)
2. MMSE≤15
3. Medicated with oral/transdermal patch anti-dementia (donepezil, rivastigmine, galantamine or memantine), alone or in combination, for a minimum period of 3 months;
4. Availability of a designated caregiver who monitors the patient's clinical situation and can collaborate in the assessment of outcomes and the provision of informed consent (ideally 8/h at least 3x/week)
5. Shared perception between the attending neurologist and family members that the drug may no longer have a therapeutic effect, has been ineffective after a therapeutic trial, or the presence of side effects possibly attributed to the drugs.

Exclusion Criteria:

1. Life expectancy presumably less than the follow-up period (6 months);
2. Unstable medical or surgical condition that can significantly interfere with the patient's overall health status;
3. Another pathology interfering with cognitive functioning (HIV, brain tumor, encephalitis, demyelinating disease);
4. Introduction of an antipsychotic drug in the last month.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
BADLS (Bristol Activities of Daily Living Scale) | 6 months
  Progression to disability (defined as a loss of 2 of 4 basic functions, or 6 of 11 instrumental functions); total score varies from 0 (totally independent) to 60 (totally dependent)
Quality of life of patients and caregivers | 6 months
  EuroQol-5D (EQ-5D); score varies from 0 to 100 using a Visual analogue scale

SECONDARY OUTCOMES:
Neuropsychiatric inventory (NPI) | 6 months
  NPI (0-144), higher scores indicating worse behavior
General Health Questionnaire 12 (caregivers) | 6 months
  score ranges from 0 to 12, with higher scores indicating increased psychological symptoms
Clinical Global Impression of Change plus Caregiver Input (CGIC-Plus) | 6 months
  The score ranges from 1 (much better) to 7 (much worse), with 4 indicating no change
Serious adverse events | 6 months
  Inpatient admission, emergency visits, antibiotic prescription, seizures, falls
Mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Verónica R Cabreira, MD, Principal Investigator — Centro Hospitalar São João (Neurology Department)
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
Upon request Supplementary data may be published along with study results.